CLINICAL TRIAL: NCT03352778
Title: Long Term Results of the Prospective Randomized Study of Intensity-modulated Radiotherapy (IMRT) Versus Two-dimensional Radiotherapy (2DRT) in Early Stage Nasopharyngeal Carcinoma (NPC) Patients
Brief Title: IMRT vs 2DRT for NPC Patients
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CCTU, Honorary clinical associate professor, Chinese University of Hong Kong
Other Study IDs: NPC031
Record Dates: First submitted 2017-11-15; First posted 2017-11-24 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: NPC

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IMRT
  Interventions: Radiation: IMRT
- 2DRT
  Interventions: Radiation: 2DRT

INTERVENTIONS:
Radiation: IMRT — 66Gy by intensity-modulated radiotherapy
  Groups: IMRT
Radiation: 2DRT — 66Gy by 2-dimensional radiotherapy
  Groups: 2DRT

SUMMARY:
Irradiation of the parotid gland with subsequent long-term xerostomia is a well-recognized complication after radiotherapy for head and neck (HAN) cancers. A number of studies have shown that IMRT could minimize the radiation dose to the parotid glands and hence the risk of developing xerostomia. The benefit of IMRT has also been demonstrated in prior dosimetric and non-randomized studies in NPC patients. In 2007, the investigators have published the prospective randomized study of IMRT versus 2DRT in early stage NPC patients. In the study, IMRT had lower incidence of observer-rated severe xerostomia, higher parotid and whole saliva flow rate, than patients in 2DRT arm at 1 year after treatment. However, there was no significant difference in patient-reported outcome, i.e. subjective xerostomia scoring, between the 2 arms. The underlying reason for the incoherent findings in terms of objective and subjective xerostomia outcome remains uncertain. One of the possible explanations for this observation could be the better parotidsparing with IMRT alone may not entirely sufficient to maintain oral cavity lubrication while the other mucin-secretory salivary gland protection is also essential. Another possible explanation for the insignificant improvement in patient-reported outcome with IMRT is the short follow-up time. Gradual recovery or improvement in various quality of life parameters was not uncommonly seen several years after definitive radiotherapy for HAN cancer patients. There is much interest in studying the long term clinical outcome, especially the treatment-related complications, for the patients who had randomized and treated in the prior presented prospective study.

In this study, the long term results, in particular the xerostomia rating will be assessed and compared in NPC patients who had participated in the prior reported prospective randomized study of IMRT vs 2DRT.

ELIGIBILITY:
Inclusion Criteria:

* The NPC patient, who had been enrolled, randomized and treated in the prior prospective randomized study of IMRT vs 2DRT.
* Regular follow-up for more than five years from the end of study intervention (i.e. IMRT or 2DRT for NPC).
* Patient is able to sign the study-specific informed consent.
* ECOG performance status 0 or 1.
* Patient is able to complete the study's questionnaire.

Exclusion Criteria:

* NPC patients who had not been randomized or allocated to the study intervention, even though had been enrolled in the prior reported study.
* Loss of regular follow-up from the end of study intervention.
* Regular follow-up for less than five years from the end of study intervention.
* Patients with known recurrent or metastatic disease.
* Patients with secondary malignancy occurred after completion of the previous study's treatment (i.e. radiotherapy).
* Active untreated infections
* Major medical or psychiatric illness

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The NPC patient, who had been enrolled, randomized and treated in the prior prospective randomized study of IMRT vs 2DRT.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
To measure QOL difference between 2DRT vs IMRT by EORTC QLQ-C30 core questionnaire. A 10-point difference of mean scores of QOL between groups were significant. | 2 years
To measure QOL difference between 2DRT vs IMRT by EORTC QLQ-H&N 35 questionnaire. A 10-point difference of mean scores of QOL between groups were significant. | 2 years
To measure difference in xerostomia score between 2DRT vs IMRT by using the xerostomia questionnaire (6-item xerostomia questionnaire. Johnson et al). A low score indicates worse xerostomia. | 2 years

SECONDARY OUTCOMES:
To measure the difference of the incidence of loco-regional recurrence between 2DRT vs IMRT. | 2 years
To measure the difference of the overall survival and progression-free survival between 2DRT vs IMRT. | 2 years
To measure the difference of numbers of 2DRT vs IMRT patients with treatment-related adverse events as assessed by RTOG/EORTC Late Radiation Morbidity Scoring Criteria. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided